CLINICAL TRIAL: NCT03484468
Title: Predictability of Corneal Flap Thickness in Lasik Using Femtosecod Laser in Comparison to Moria Microkeratome
Brief Title: Femtosecond Laser Versus Microkeratome in Creating Corneal Flaps in LASIK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gerges Fargalla, Medicin Baccalaureus et Baccalaureus Chirurgi, Assiut University
Other Study IDs: femtosecond_vs_microkeratome
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Femtosecond Laser in Comparison to Moria Microkeratome in Creating Corneal Flaps
Keywords: lasik; flap_thickness; femtosecond; laser; moria; microkeratome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- femtosecond_laser: participants had there lasik corneal flap creation using femtosecond laser
  Interventions: Device: anterior segment Ocular Coherence Tomography
- moria_microkeratome: participants had there lasik corneal flap creation using moria microkeratome
  Interventions: Device: anterior segment Ocular Coherence Tomography

INTERVENTIONS:
Device: anterior segment Ocular Coherence Tomography — anterior segment OCT (Ocular Coherence Tomography) a device shows imaging of anterior segment of the eye and able to show corneal layers and measures its thickness.

SUMMARY:
Since the cornea is the main responsible for the refraction of the eye, as its refractive power is greater than 70% of the total refraction of the eye, so modification of its refractive properties are used to change the optical system of the eye. Hence, laser-assisted in situ keratomileusis has become the most commonly procedure used to correct the refractive errors of the eye. The most important step in laser-assisted in situ keratomileusis is the creation of the corneal flap, which its thickness may judge the whole outcome of the surgery . So trying to minimize the variation in the thickness of the resultant flap in comparison to what planned flap thickness preoperatively become our target.

DETAILED DESCRIPTION:
As laser-assisted in situ keratomileusis procedure started to use automated microkeratomes in creating corneal flaps since 1989, and science go on until United states Food and Drug Administration approved the IntraLase laser for flap creation in January 2000 femtosecond lasers work by emitting light pulses of short duration (10-15 s) at 1053 nm wavelength that cause photodisruption of the tissue with minimum collateral damage . This enables no blade incisions to be performed within the tissue at various patterns and depth with high precision.

Aim of the work To evaluate and compare the variation in corneal flap thickness created from use of a femtosecond laser and a MORIA microkeratome when making a 110-µm- and 90- µm thick corneal flap and to identify the potential factors that affect corneal flap thickness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 year
* Preoperative spherical refraction of -2.00 to -10.00D.
* Refractive cylinder of less than -3.00D.
* A stable refractive state for 2 years.
* An intraocular pressure (IOP) of <22 mm Hg.

Exclusion Criteria:

* A history of any systemic autoimmune disease.
* A history of diabetes.
* Other ophthalmic disorders.
* A history of ocular trauma and surgical history.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: population attending specialized eye centers
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
corneal flap thickness | 7 days
  measuring the corneal flap thickness in nanometers postoperatively by anterior segment OCT

SECONDARY OUTCOMES:
uncorrected visual acuity | 7 days
  identifying uncorrected visual acuity postoperatively
best corrected visual acuity | 7 days
  identifying best corrected visual acuity postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: GERGES F. YOUNAN, M.B.B.CH., Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang J, Zhang SS, Yu Q, Wu JX, Lian JC. Comparison of corneal flap thickness using a FS200 femtosecond laser and a moria SBK microkeratome. Int J Ophthalmol. 2014 Apr 18;7(2):273-7. doi: 10.3980/j.issn.2222-3959.2014.02.14. eCollection 2014. PMID 24790869
- [Result] F.A.Guarnieri(ed.), Introduction, Corneal Biomechanics and Refractive Surgery, © Springer Science+Business Media New York 2015 ; 1: 1
- [Result] Solomon KD, Fernandez de Castro LE, Sandoval HP, Biber JM, Groat B, Neff KD, Ying MS, French JW, Donnenfeld ED, Lindstrom RL; Joint LASIK Study Task Force. LASIK world literature review: quality of life and patient satisfaction. Ophthalmology. 2009 Apr;116(4):691-701. doi: 10.1016/j.ophtha.2008.12.037. PMID 19344821
- [Result] Sugar A, Rapuano CJ, Culbertson WW, Huang D, Varley GA, Agapitos PJ, de Luise VP, Koch DD. Laser in situ keratomileusis for myopia and astigmatism: safety and efficacy: a report by the American Academy of Ophthalmology. Ophthalmology. 2002 Jan;109(1):175-87. doi: 10.1016/s0161-6420(01)00966-6. PMID 11772601
- [Result] Hsu SY, Chen HY, Chung CP. Analysis of actual corneal flap thickness and confounding factors between first and second operated eyes. Ophthalmic Surg Lasers Imaging. 2009 Sep-Oct;40(5):448-52. doi: 10.3928/15428877-20090901-02. PMID 19772267
- [Result] Ortiz D, Alio JL, Pinero D. Measurement of corneal curvature change after mechanical laser in situ keratomileusis flap creation and femtosecond laser flap creation. J Cataract Refract Surg. 2008 Feb;34(2):238-42. doi: 10.1016/j.jcrs.2007.09.023. PMID 18242446
- [Result] Reinstein DZ, Archer TJ, Gobbe M. The history of LASIK. J Refract Surg. 2012 Apr;28(4):291-8. doi: 10.3928/1081597X-20120229-01. PMID 22496438
- [Result] Soong HK, Malta JB. Femtosecond lasers in ophthalmology. Am J Ophthalmol. 2009 Feb;147(2):189-197.e2. doi: 10.1016/j.ajo.2008.08.026. Epub 2008 Oct 18. PMID 18930447
- [Result] Marino GK, Santhiago MR, Wilson SE. Femtosecond Lasers and Corneal Surgical Procedures. Asia Pac J Ophthalmol (Phila). 2017 Sep-Oct;6(5):456-464. doi: 10.22608/APO.2017163. Epub 2017 Jul 31. PMID 28780779
- [Result] Ratkay-Traub I, Ferincz IE, Juhasz T, Kurtz RM, Krueger RR. First clinical results with the femtosecond neodynium-glass laser in refractive surgery. J Refract Surg. 2003 Mar-Apr;19(2):94-103. doi: 10.3928/1081-597X-20030301-03. PMID 12701713